CLINICAL TRIAL: NCT05090891
Title: A Phase 2, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Efficacy, Safety, and Tolerability of INCB000928 in Participants With Fibrodysplasia Ossificans Progressiva
Brief Title: To Assess the Efficacy, Safety, and Tolerability of INCB000928 in Participants With Fibrodysplasia Ossificans Progressiva
Acronym: Progress
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Incyte Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: INCB 00928-201; 2023-504129-38-00 (Registry Identifier: EU CT Number); 2021-002286-17 (EudraCT Number)
Record Dates: First submitted 2021-10-08; First posted 2021-10-25 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-12

CONDITIONS: Fibrodysplasia Ossificans Progressiva (FOP)
Keywords: fibrodysplasia ossificans progressiva (FOP); heterotopic ossification
MeSH Terms: conditions — Myositis Ossificans; Ossification, Heterotopic

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Cohort 1 (Experimental): Participants (≥ 12 years of age) will receive INCB000928 or placebo as defined in the protocol for 24 weeks (double-blind period). Participants who complete the double-blind period will continue into open-label extension period for an additional 292 weeks.
  Interventions: Drug: INCB000928; Drug: Placebo
- Cohort 2 (Experimental): Participants (6 to < 12 years of age) will receive INCB000928 or placebo as defined in the protocol for 24 weeks (double-blind period). Participants who complete the double-blind period will continue into open-label extension period for an additional 292 weeks.
  Interventions: Drug: INCB000928; Drug: Placebo
- Cohort 3 (Experimental): Participants (2 to < 6 years of age) will receive INCB000928 or placebo as defined in the protocol for 24 weeks (double-blind period). Participants who complete the double-blind period will continue into open-label extension period for an additional 292 weeks.
  Interventions: Drug: INCB000928; Drug: Placebo

INTERVENTIONS:
Drug: INCB000928 — INCBG000928 will be administered QD orally.
  Other Names: zilurgisertib
Drug: Placebo — Placebo will be administered QD orally.

SUMMARY:
This Phase 2, Randomized, Double-Blind, Placebo-Controlled Study is intended to evaluate the Efficacy, Safety, and Tolerability and PK of INCB000928 administered to participants with a clinical diagnosis of fibrodysplasia ossificans progressiva (FOP).

ELIGIBILITY:
Inclusion Criteria:

* Female and male participants:

  * Cohort 1: ≥ 12 years of age.
  * Cohort 2: 6 to < 12 years of age.
  * Cohort 3: 2 to < 6 years of age (after eDMC review of interim data from Cohort 2).
* Clinical diagnosis of FOP.
* Willingness to avoid pregnancy or fathering children based on the criteria below.
* Willing and able to undergo low-dose WBCT (excluding the head) imaging without requiring intubation.
* Further inclusion criteria apply.

Exclusion Criteria:

* Pregnant or breast-feeding.
* CAJIS score ≥ 24.
* FOP disease severity that in the investigator's opinion precludes participation.
* Any clinically significant medical condition other than FOP that would, in the investigator's judgment, interfere with full participation in the study, pose a significant risk to the participant, or interfere with interpretation of study data.
* Chronic or current active infectious disease requiring systemic antibiotic, antifungal, or antiviral treatment.
* HIV, HBV, or HCV infection. Note:
* Further exclusion criteria apply.

Ages: 2 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 98 (Estimated)
Dates: Start 2022-05-05 (Actual); Primary Completion 2027-07-30 (Estimated); Study Completion 2033-01-20 (Estimated)

PRIMARY OUTCOMES:
Double Blind Period: Occurrence of new heterotopic ossification (HO) lesions from baseline | Week 24
  HO will be assessed by low dose whole-body computed tomography (WBCT) (excluding the head) compared to baseline during the double-blind period.

SECONDARY OUTCOMES:
Double Blind Period: Number of new HO lesions from baseline | Week 24
  HO will be assessed by low dose whole-body computed tomography (WBCT) (excluding the head) compared to baseline during the double-blind period.
Double Blind Period: Total volume of new HO lesions from baseline | Week 24
  HO will be assessed by low dose whole-body computed tomography (WBCT) (excluding the head) compared to baseline during the double-blind period.
Double Blind Period: Change in the total volume of all HO lesions from baseline | Week 24
  HO will be assessed by low dose whole-body computed tomography (WBCT) (excluding the head) compared to baseline during the double-blind period.
Double Blind Period: Number of new flares from baseline | Week 24
  Based on Fibrodysplasia Ossificans Progressiva - Patient RepOrted syMPtoms Tool (FOP-PROMPT).
Number of Participants with Treatment Emergent Adverse Events (TEAE) | Up to 316 weeks
  Defined as any adverse event either reported for the first time or worsening of a pre-existing event after first dose of study drug.
Open-Label Extension: Occurrence of new HO lesions from Week 24 | Week 48
  HO will be assessed by low dose whole-body computed tomography (WBCT) (excluding the head) from Week 24 to Week 48 compared to baseline to Week 24 in participants randomized to placebo during the DB period.
Open-Label Extension: Number of new HO lesions from Week 24 | Week 48
  HO will be assessed by low dose whole-body computed tomography (WBCT) (excluding the head) from Week 24 to Week 48 compared to baseline to Week 24 in participants randomized to placebo during the DB period.
Open-Label Extension: Total volume of new HO lesions from Week 24 | Week 48
  HO will be assessed by low dose whole-body computed tomography (WBCT) (excluding the head) from Week 24 to Week 48 compared to baseline to Week 24 in participants randomized to placebo during the DB period.
Open-Label Extension: Change in the total volume of all HO lesions from Week 24 | Week 48
  HO will be assessed by low dose whole-body computed tomography (WBCT) (excluding the head) from Week 24 to Week 48 compared to baseline to Week 24 in participants randomized to placebo during the DB period.
Open-Label Extension: Number of new flares from Week 24 | Week 48
  Based on Fibrodysplasia Ossificans Progressiva - Patient RepOrted syMPtoms Tool (FOP-PROMPT) from Week 24 to Week 48 compared to baseline to Week 24 in participants randomized to placebo during the DB period.
Pharmacokinetics Parameter: Cmax of INCB000928 | Baseline, Weeks 12, 24, 48 and 76
  Maximum observed concentration.
Pharmacokinetics Parameter: Tmax of INCB000928 | Baseline, Weeks 12, 24, 48 and 76
  Time to maximum concentration.
Pharmacokinetics Parameter: Cmin of INCB000928 | Baseline, Weeks 12, 24, 48 and 76
  Minimum observed concentration.
Pharmacokinetics Parameter: AUCt of INCB000928 | Baseline, Weeks 12, 24, 48 and 76
  Area under the plasma concentration-time curve from time 0 to the last quantifiable measurable plasma concentration

CONTACTS AND LOCATIONS:
Overall Officials: Amanda McBride, MD, Study Director — Incyte Corporation
Locations (27):
- United States (4):
  - University of California San Francisco Medical Center, San Francisco, California
  - Mayo Clinic Rochester, Rochester, Minnesota
  - Children'S Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Penn Medicine - Perelman Center For Advanced Medicine, Philadelphia, Pennsylvania
- Hospital Italiano de Buenos Aires, Ciudad Autonoma Buenos Aires, Argentina
- Australia (2):
  - Royal North Shore Hospital, St Leonards, New South Wales
  - Murdoch Children'S Research Institute, Parkville, Victoria
- Albert Einstein Israelite Hospital, São Paulo, Brazil
- University Health Network Toronto General Hospital, Toronto, Ontario, Canada
- Centro de Estudios Reumatologicos, Santiago, Chile
- China (4):
  - Beijing Childrens Hospital Capital Medical University, Beijing
  - Tongji Hospital of Tongji University, Shanghai
  - Shanghai Childrens Medical Center, Shanghai
  - Childrens Hospital of Fudan University, Shanghai
- France (2):
  - Ap-Hp Hopital Lariboisiere, Paris
  - Hopital Necker-Enfants Malades, Paris
- Uniklinik Koln, Cologne, Germany
- Italy (2):
  - Ospedale Pediatrico G. Gaslini, Genova
  - Policlinico Universitario Agostino Gemelli Universita Cattolica Del Sacro Cuore, Rome
- Instituto Nacional de Rehabilitacion Luis Guillermo Ibarra, Tlalpan, Mexico
- Amsterdam Umc - Vu Medisch Centrum (Vumc), Amsterdam, Netherlands
- Starship Childrens Hospital, Auckland, New Zealand
- Groote Schuur Hospital Radiation Oncology, Cape Town, South Africa
- Seoul National University Hospital, Seoul, South Korea
- Hospital Universitario Ramon Y Cajal, Madrid, Spain
- United Kingdom (2):
  - Royal Manchester Childrens Hospital - Department of Paediatric Endocrinology, Manchester
  - Royal National Orthopaedic Hospital, Stanmore

IPD SHARING:
Plan to Share IPD: Yes
Incyte shares data with qualified external researchers after a research proposal is submitted. These requests are reviewed and approved by a review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
Supporting Information: Study Protocol, SAP
Time Frame: Data will be shared after the primary publication or 2 years after the study has ended for market authorized products and indications.
Access Criteria: Data from eligible studies will be shared with qualified researchers according to the criteria and process described in the Data Sharing section of the www.incyteclinicaltrials.com website. For approved requests, the researchers will be granted access to anonymized data under the terms of a data sharing agreement.
URL: https://www.incyte.com/our-company/compliance-and-transparency

REFERENCES:
- [Derived] Yang YO, Fang Y, Wang P, Liu X, Getsy J, Rockich K. Effects of Renal and Hepatic Impairment on the Pharmacokinetics of Zilurgisertib. Br J Clin Pharmacol. 2025 Dec 8. doi: 10.1002/bcp.70372. Online ahead of print. PMID 41360500
- See also: To Assess the Efficacy, Safety, and Tolerability of INCB000928 in Participants With Fibrodysplasia Ossificans Progressiva (Progress) — https://www.incyteclinicaltrials.com/study/?id=INCB%2000928-201&SearchTerm=INCB%2000928-201&Latitude=&Longitude=&LocationName=&conditions=&Status=&phases=&AgeRanges=&gender=&StudyTypes=&AttachmentTypes=&MileRadius=100&PageIndex=0&PageSize=10&SortField=&SortOrder=&hasResults=